CLINICAL TRIAL: NCT00656669
Title: An Exploratory Study of the Biological and Clinical Activity of Sunitinib Malate as a Component of Neoadjuvant Therapy for Breast Cancer
Brief Title: Exploratory Study of Sunitinib Malate as a Component of Neoadjuvant Therapy for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Kathy Miller, Professor of Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0802-15/1011003564; IUCRO-0215
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: newly diagnosed breast cancer; neoadjuvant therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Sunitinib; Paclitaxel; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): The study will be conducted in 3 sequential treatment segments.
  Interventions: Drug: sunitinib alone; Drug: sunitinib plus paclitaxel; Drug: doxorubicin and cyclophosphamide

INTERVENTIONS:
Drug: sunitinib alone — sunitinib alone (segment 1): During the first segment, patients will receive single-agent sunitinib for 2 weeks.
Drug: sunitinib plus paclitaxel — sunitinib plus paclitaxel (Segment 2): Following Segment 1, patients will begin the second segment, 4 cycles (16 weeks) of neoadjuvant treatment with the combination of sunitinib and paclitaxel.
Drug: doxorubicin and cyclophosphamide — doxorubicin and cyclophosphamide (Segment 3): Following Segment 2, patients will receive 4 cycles (8 weeks) of neoadjuvant treatment with AC.

SUMMARY:
The combination of paclitaxel, doxorubicin, and cyclophosphamide is a standard neoadjuvant (given before surgery) treatment for patients that have either inoperable or operable breast cancer. This treatment can help shrink the tumors so they can be removed to help prevent the cancer from spreading to other parts of the body. This study is being done to test the impact of adding sunitinib as a single-agent (Segment 1), followed by sunitinib plus paclitaxel (Segment 2), followed by doxorubicin and cyclophosphamide (Segment 3). We hope the addition of sunitinib will make the treatment more effective, but we don't know if this is true.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically-confirmed adenocarcinoma of the breast with operable or inoperable stage 1c (primary tumor > 1.0 cm), II or III disease.
2. Measurable disease by physical examinations or diagnostic breast imaging (mammography, ultrasonography or MR).
3. Pre-treatment core or incisional biopsy. Patients may not have had definitive primary surgery.
4. Male or female, 18 years of age or older.
5. ECOG performance status 0 or 1.
6. Adequate organ function as defined in the protocol.

Exclusion Criteria:

1. Prior radiation therapy, cytotoxic therapy or systemic therapy for breast cancer. Prior use of tamoxifen or raloxifene as chemoprevention is allowed but must be discontinued prior to study entry.
2. Metastatic (Stage IV) breast cancer
3. Patients who have had only a pre-treatment fine needle aspiration (FNA) are excluded.
4. Current therapeutic treatment on another clinical trial with an investigational agent.
5. Any of the following within the 6 months prior to starting study treatment: -myocardial infarction -severe/unstable angina -coronary/peripheral artery bypass graft -congestive heart failure -cerebrovascular accident including transient ischemic attack -pulmonary embolus
6. Ongoing cardiac dysrhythmias of NCI CTCAE grade >=2, atrial fibrillation of any grade, or QTc interval >450 msec for males or >470 msec for females.
7. Hypertension that cannot be controlled by medications.
8. Current treatment with therapeutic doses of any anti-coagulant. Prophylactic use of anticoagulants is allowed.
9. Known human immunodeficiency virus (HIV) infection.
10. Pregnancy or breastfeeding. All female patients with reproductive potential must have a negative pregnancy test prior to first day of study medication.
11. Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Please note that one patient discontinued due to an Adverse Event after completing Segment 2 (Paclitaxel/Sunitinib), but before starting Segment 3 adriamycin & cyclophosphamide (AC).
Groups:
- Segment Information: This is an exploratory phase 2 and biomarker clinical trial of sunitinib in the neoadjuvant setting for the treatment of breast cancer. The study will be conducted in 3 sequential treatment segments. During the first segment, patients will receive single-agent sunitinib for 2 weeks for the purpose of biomarker and IFP evaluation. Patients will then begin the second segment, 4 cycles (16 weeks) of neoadjuvant treatment with the combination of sunitinib and paclitaxel. Sunitinib will be discontinued after Cycle 5 Day 21. The third segment will include 4 cycles (8 weeks) of neoadjuvant treatment with AC followed by surgical resection and determination of pathological response.
Period: Single Agent Sunitinib (Cycle 1)
Arm/Group | Segment Information
Started | 23
Completed | 23
Not Completed | 0
Period: Paclitaxel/Sunitinib (Cycles 2-5)
Arm/Group | Segment Information
Started | 23
Completed | 17
Not Completed | 6
Not completed — Adverse Event | 4
Not completed — Physician Decision | 2
Period: AC (Cycles 6-9)
Arm/Group | Segment Information
Started | 17
Completed | 15
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Did not start segment 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: These patients are for the patients who were into the trial.
Arm/Group | Overall Study
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.3 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Interstitial Fluid Pressure (IFP) Induced by Sunitinib Monotherapy
Description: Participants had their tumor IFP measured at baseline, after sunitinib monotherapy (segment 1) and after sunitinib+paclitaxel (segment 2). This outcome measure is the difference of the mean value from the end of segment 1 (sunitinib monotherapy) and the mean baseline value.
Time Frame: baseline through end of segment 1 (2 weeks)
Population: All patients that had both measures at baseline and endpoint in the sunitinib monotherapy segment
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Sunitinib Monotherapy: Patients who completed the Sunitinib monotherapy segment
Arm/Group | Sunitinib Monotherapy
Number analyzed (Participants) | 19
mm Hg | 14.0 (12.4)
Statistical Analysis 1: Comparison: Sunitinib Monotherapy; From Taghian et al., we used a mean IFP of 6.5 at baseline and a standard deviation of 6.1. We would like to detect a 50% reduction of IFP (to 3.25 mmHg) with sunitinib monotherapy, so the effect size would be 3.25/6.1=0.53. A two-sided paired t-test has 80% power to detect an effect size of .53 and level of significance .05 when the sample size is 30 patients; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided; This is a paired t-test to compare baseline IFP to IFP after completion of sunitinib monotherapy

2. Secondary Outcome: Change in Interstitial Fluid Pressure (IFP) Induced by Paclitaxel Plus Sunitinib After Sunitinib Monotherapy
Description: Participants had their tumor IFP measured at baseline, after sunitinib monotherapy (segment 1) and after sunitinib+paclitaxel (segment 2). This outcome measure is the difference of the mean value from the end of segment 2 (paclitaxel/sunitinib therapy through cycle 5) and end of segment 1 (sunitinib monotherapy) mean value.
Time Frame: end of cycle 1 (sunitinib monotherapy) to end of cycle 5 (paclitaxel/sunitinib therapy) (112 days)
Population: All patients in the paclitaxel plus sunitinib segment
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Paclitaxel Plus Sunitinib: Patients who finished the paclitaxel plus sunitinib segment
Arm/Group | Paclitaxel Plus Sunitinib
Number analyzed (Participants) | 6
mm Hg | 1.7 (15.2)
Statistical Analysis 1: Comparison: Paclitaxel Plus Sunitinib; Test type: Superiority or Other; p = 0.7963, t-test, 2 sided — a priori threshold of <0.05; This is a paired t-test to compare baseline IFP to IFP after completion of paxlitaxel+sunitinib treatment

3. Secondary Outcome: Pathological Complete Response (pCR) Rate for Patients Treated With Sunitinib/Paclitaxel Followed by AC as Neoadjuvant Therapy for Breast Cancer
Time Frame: screening through surgery
Population: All patients who had surgery.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- AC Dosing: Patients who finished the AC dosing segment
Arm/Group | AC Dosing
Number analyzed (Participants) | 15
percentage of participants | 53.3 [26.6 to 78.7]

4. Secondary Outcome: To Evaluate the Safety of Paclitaxel Plus Sunitinib When Given in Combination as Neoadjuvant Therapy
Description: This measure determines the number of patients who had Grade 3/4 Adverse Events that were related to treatment while the patient was on paclitaxel plus sunitinib.
Time Frame: end of cycle 1 (sunitinib monotherapy) to end of cycle 5 (paclitaxel/sunitinib therapy)
Population: All patients who were on paclitaxel plus sunitinib.
Measure: Number; unit: participants
Groups:
- Paclitaxel Plus Sunitinib: Patients who were in the paclitaxel plus sunitinib segment
Arm/Group | Paclitaxel Plus Sunitinib
Number analyzed (Participants) | 23
participants | 11

ADVERSE EVENTS:
Time Frame: Cycles 1 through 9 of treatment
Groups:
- Single Agent Sunitinib: Single-agent sunitinib for 2 weeks for the purpose of biomarker and IFP evaluation.
- Paclitaxel/Sunitinib: 4 cycles (16 weeks) of neoadjuvant treatment with the combination of sunitinib and paclitaxel.
- AC Dosing: 4 cycles (8 weeks) of neoadjuvant treatment with AC.
Arm/Group | Single Agent Sunitinib | Paclitaxel/Sunitinib | AC Dosing
Serious Adverse Events (participants affected / at risk) | 0/23 | 2/23 | 2/16
Other Adverse Events (participants affected / at risk) | 20/23 | 22/23 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Agent Sunitinib (N=23) | Paclitaxel/Sunitinib (N=23) | AC Dosing (N=16)
LEFT VENTRICULAR SYSTOLIC DYSFUNCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
BILIRUBIN (HYPERBILIRUBINEMIA) (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
INFECTION (DOCUMENTED CLINICALLY OR MICROBIOLOGICALLY) WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Investigations) | 0 (0) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (FEVER OF UNKNOWN ORIGIN WITHOUT CLINICALLY OR MICROBIOLOGICALLY DOCUMENTED INFE (Investigations) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Agent Sunitinib (N=23) | Paclitaxel/Sunitinib (N=23) | AC Dosing (N=16)
DERMAL CHANGE LYMPHEDEMA, PHLEBOLYMPHEDEMA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (2)
LEFT VENTRICULAR SYSTOLIC DYSFUNCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
VENTRICULAR ARRHYTHMIA - VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
DRY EYE SYNDROME (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
OCULAR/VISUAL - OTHER (SPECIFY, __) (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
VISION-BLURRED VISION (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (5)
DIARRHEA (Gastrointestinal disorders) | 6 (6) | 13 (17) | 2 (2)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 5 (5) | 12 (21) | 3 (3)
HEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) - ORAL CAVITY (Gastrointestinal disorders) | 6 (6) | 8 (11) | 3 (3)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) - ORAL CAVITY (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) - STOMACH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 8 (8) | 10 (16) | 6 (10)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 11 (12) | 13 (19) | 4 (4)
VOMITING (Gastrointestinal disorders) | 5 (5) | 3 (4) | 5 (7)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 7 (7) | 15 (22) | 7 (11)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 2 (3) | 0 (0) | 3 (3)
PAIN - ABDOMEN NOS (General disorders) | 0 (0) | 3 (3) | 1 (1)
PAIN - BACK (General disorders) | 0 (0) | 2 (3) | 3 (3)
PAIN - BREAST (General disorders) | 2 (2) | 2 (3) | 0 (0)
PAIN - CARDIAC/HEART (General disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN - CHEST/THORAX NOS (General disorders) | 0 (0) | 1 (1) | 1 (1)
PAIN - EXTREMITY-LIMB (General disorders) | 0 (0) | 3 (5) | 1 (1)
PAIN - HEAD/HEADACHE (General disorders) | 3 (3) | 2 (2) | 2 (2)
PAIN - JOINT (General disorders) | 1 (1) | 4 (4) | 3 (4)
PAIN - MUSCLE (General disorders) | 1 (1) | 5 (6) | 2 (2)
PAIN - OTHER (SPECIFY, __) (General disorders) | 0 (0) | 2 (4) | 0 (0)
PAIN - STOMACH (General disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN - THROAT/PHARYNX/LARYNX (General disorders) | 1 (1) | 1 (3) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - PARANASAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - SINUS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - SKIN (CELLULITIS) (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - UPPER AIRWAY NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTION WITH UNKNOWN ANC - URINARY TRACT NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
BURN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 0 (0) | 1 (1) | 1 (1)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 0 (0) | 1 (1) | 1 (1)
HEMOGLOBIN (Investigations) | 0 (0) | 0 (0) | 1 (3)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Investigations) | 0 (0) | 10 (14) | 1 (1)
PLATELETS (Investigations) | 0 (0) | 4 (4) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 5 (6) | 12 (18) | 8 (9)
NEUROPATHY: SENSORY (Nervous system disorders) | 4 (4) | 11 (17) | 1 (1)
INSOMNIA (Psychiatric disorders) | 2 (2) | 8 (9) | 2 (2)
MOOD ALTERATION - ANXIETY (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0)
MOOD ALTERATION - DEPRESSION (Psychiatric disorders) | 1 (1) | 4 (4) | 2 (2)
HOT FLASHES/FLUSHES (Reproductive system and breast disorders) | 0 (0) | 5 (5) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 10 (14) | 3 (3)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 9 (10) | 2 (2)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY - NOSE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 0 (0)
PULMONARY/UPPER RESPIRATORY - OTHER (SPECIFY, __) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 1 (1) | 18 (23) | 2 (2)
HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
HYPOPIGMENTATION (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (9) | 1 (1)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5) | 0 (0)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 3 (4) | 5 (7) | 3 (3)
RASH: HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (10) | 2 (2)
HYPERTENSION (Vascular disorders) | 4 (4) | 7 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes